CLINICAL TRIAL: NCT04641598
Title: The Effect of Menstrual Phase Endometrial Scratch on Intrauterine Insemination Cycle Outcomes and Participant Acceptability
Brief Title: Menstrual Phase Endometrial Scratch in IUI Cycles
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment is low and interim analysis demonstrated no difference in outcomes.
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Emily Evans-Hoeker, Principal Investigator, Physician, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-20-1017
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Fertility Disorders; Fertility Issues
Keywords: infertility; insemination
MeSH Terms: conditions — Infertility | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are randomized to endometrial scratch or "sham" procedure (speculum insertion but no endometrial scratch)
Who Masked: Participant
Masking Description: Participants are not made aware of which arm they are randomized to until after the cycle outcome has been determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endometrial scratch (Experimental): A speculum will be inserted into the vagina and the cervix cleansed with betadine (or alternative if allergy). The cervix will be grasped with a single tooth tenaculum and an endometrial biopsy pipelle inserted into the uterine cavity to the depth of the uterine fundus. Suction will be applied and the pipelle will be completely withdrawn in a single pass. All instruments will be removed from the vagina after hemostasis is ensured.
  Interventions: Procedure: Endometrial Scratch
- Sham procedure (Sham Comparator): A speculum will be inserted into the vagina and the cervix cleansed with betadine (or alternative if allergy). The motions of grasping the cervix with a single tooth tenaculum and inserting the biopsy pipelle will be simulated, but not actually performed. All instruments will then be removed from the vagina.
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Procedure: Endometrial Scratch — An endometrial biopsy pipelle will be used to create endometrial injury in the form of a "scratch".
  Other Names: Endometrial injury
  Arms: Endometrial scratch
Procedure: Sham procedure — Motions of performing an endometrial scratch will be performed including speculum placement and cervix cleansing, however, placement of the tenaculum and the endometrial scratch will not be performed.
  Other Names: Sham
  Arms: Sham procedure

SUMMARY:
Patients undergoing treatment with intrauterine insemination (IUI) will be randomized to receive an endometrial scratch or sham procedure during the menstrual phase of the treatment cycle.

DETAILED DESCRIPTION:
Infertility is a common issue faced by many couples throughout the United States. There are multiple fertility treatment options, including in vitro fertilization (IVF) and intrauterine insemination (IUI). Additionally, methods such as endometrial scratch (a modified endometrial biopsy) have been postulated to increase success rate. This prospective, randomized control trial will assess whether performing an endometrial scratch improves cycle outcomes and decreases time to pregnancy following IUI. Each patient will be randomly assigned to receive either an endometrial scratch or undergo a "sham" procedure (speculum insertion but no scratch) during the menstrual phase of the IUI cycle.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing intrauterine insemination procedures between the ages of 18 and 37 who have undergone a complete fertility work up (tubal, uterine, hormonal and sperm assessments) and do not have a current tubal or uterine factor infertility or severe male factor (expected to have < 10 million total motile sperm on IUI sample) unless using donor sperm.

Exclusion Criteria:

* age < 18 or > 37, expectation (prior to randomization) of < 10 million total motile sperm on IUI sample, tubal factor, uterine factor, incomplete fertility work up.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants are all undergoing intrauterine insemination and thus must have a uterus. This definition is based on anatomy rather than gender identity.
Enrollment: 57 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | Within one month from study randomization.
  Obtaining a positive pregnancy test (urine or serum) at the conclusion of the treatment cycle in which the scratch was performed.

SECONDARY OUTCOMES:
Time to conception | To be assessed within 6 months of randomization.
  The amount of time between study randomization and positive pregnancy test.
Participants perceived acceptability | The survey assessing this outcome is completed by the participant on the day of the study procedure.
  Participants rating of acceptability of the study procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Hoeker, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic Reproductive Medicine and Fertility, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to make IPD available to other researchers.

REFERENCES:
- [Background] Wadhwa L, Pritam A, Gupta T, Gupta S, Arora S, Chandoke R. Effect of endometrial biopsy on intrauterine insemination outcome in controlled ovarian stimulation cycle. J Hum Reprod Sci. 2015 Jul-Sep;8(3):151-8. doi: 10.4103/0974-1208.165144. PMID 26538858